CLINICAL TRIAL: NCT03914599
Title: Protective Genetic Factors Against Neurological Diseases
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Jun Li, Chair and Professor of Department of Neurology, Wayne State University
Other Study IDs: 08675309
Record Dates: First submitted 2019-04-01; First posted 2019-04-16 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Neurological Disorder; Healthy Control
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — All research participants, including healthy control volunteers, will be asked to give their blood samples once they are enrolled into the study. Their DNA will be extracted from the blood samples and stored in the freezers at the Integrative Biosciences Center in Detroit, MI. All samples stored in the Biobank at iBIO will be frozen and kept for an indefinite amount of time. The participant cannot obtain or access the stored samples in the future nor will participants have access to information or test results obtained from their personal samples because personal identifiers will be removed from the samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurological Disorder: For all neurological disorder participants an electromyography (EMG) study will be done to determine nerve conduction speed, and a blood draw will be completed for genetic (DNA) testing. Motor measures, cognitive measures and surveys will be completed to assess walking and brain processing speed. Four optional assessments will be offered and only completed if the participant consents to them and include: optical coherence tomography (pictures of the back of the eye), visual evoked potential (to evaluate the nerve pathways of the eye), brain MRI, and skin biopsy. For participants with a diagnosis of Charcot Marie Tooth (CMT) disease, they will have an additional Neuropathy Score to assess disease severity.
- Healthy Control: An electromyography (EMG) study will be done to determine nerve conduction speed, and a blood draw will be completed for genetic (DNA) testing. Motor measures, cognitive measures and surveys will be completed to assess walking and brain processing speed. Four optional assessments will be offered and only completed if the participant consents to them and include: optical coherence tomography (pictures of the back of the eye), visual evoked potential (to evaluate the nerve pathways of the eye), brain MRI, and skin biopsy.

SUMMARY:
NIH Precision Medicine Initiative, started in May 2018, will enroll one million people through an online portal. It hopes to identify genetic variants affecting a variety of human phenotypic outcomes. A giant set of data like this may enable an association of genetic variants with a certain phenotype. However, the association is often compromised due to the collection of phenotypic data that is not well controlled or standardized creating "noisy" data. These phenotypic "noises" can be largely eliminated in clinical studies with stringent criteria and standardization of outcome measurements.

In this study, by looking mainly at genetic information and nerve conduction speed, we hope to eliminate the extra "noises" in the data set. Eliminating the extra "noises" should allow us to be able to determine if there are genetic differences between neurological disorders and healthy controls, and if these genetic differences can be attributed to the speed of the nerve conduction.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a neurological disorder - Inherited Peripheral Neuropathy, Charcot Marie Tooth, Multiple Sclerosis, or Parkinson's Disease
2. Healthy volunteers with no history of medical conditions known to afflict the nervous system will be recruited as normal controls.
3. Age 18-100 (Inclusive)
4. Able to undergo MRI
5. Medically Stable

Exclusion Criteria:

1. Any subject unwilling to undergo genetic testing (DNA sampling)
2. Any subjects with history of peripheral nerve diseases or conditions known to affect the CNS, such as diabetes, stroke, thyroid disease, chemotherapy, renal failure, etc.

Note: This study holds no additional risk for pregnant women and they will not be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurology clinic for participants with a diagnosis of a neurological disorder and fliers will be posted for healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Association of human genetic variants with the fastest conduction speed in normal controls | 5 years
  nerve conduction velocity as measured by electromyogram machine
The cluster of genetic variants associated with the fastest conduction velocity in normal controls versus those altered in patients with neurological diseases will be characterized | 5 years
  nerve conduction velocity and neurological disability scores as assessed by Visser Neuropathy Score ranging from 0-68 with higher score indicating more severe disabilities.
To test if the genetic variants associated with the fastest CV in the PNS protect some patients with CMT1A from developing severe disabilities | 5 years
  neurological disability scores as assessed by Visser Neuropathy Score ranging from 0-68 with higher score indicating more severe disabilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States